CLINICAL TRIAL: NCT06189534
Title: Cognitive Behavior Therapy for Social Media Addiction, Insomnia, and Family Relationship Among Individuals With Social Media Addiction: A Randomized Control Tria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Dr Qaiser Abbas [Assistant Professor Clinical Psychology], Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GovernmentCUF.
Record Dates: First submitted 2023-11-29; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Behavior Therapy for Social Media Addiction
Keywords: Social media addiction; Insomnia; Family bonding; Cognitive behavioral therapy
MeSH Terms: conditions — Internet Addiction Disorder; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: It was an experimental pre-test post-test research design which investigated the social media addiction, insomnia poor family bonding and effectiveness of cognitive behavior interventions in managing social media addiction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms of the study (Experimental): Experimental group : participants in experimental group will receive 8-10 sessions of intervention in overall the course of study.
  Interventions: Behavioral: Cognitive behavioral therapy
- Control group (No Intervention): Control group: participants in control group will not receive any sessions of intervention.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy-based interventions were used to manage social media addiction and; to address associated problems with it. Psychoeducation, problem conceptualization, cognitive distortions and belief identification,Time management,Stress and distress management, Emotional and beliefs modification,Priority and Goal setting, Problem solving skills, Social skill training, Emotional and behavioral activation and Relapse prevention are techniques that will be used in the intervention.
  Arms: Arms of the study

SUMMARY:
Objectives This study is designed to investigate the following objectives To manage the social media addiction in order to improve lifestyle, attitude and family relations of the individuals and explore related psychological problems which can arise because of this addiction.

To explore the effectiveness of cognitive behaviour therapy (CBT) in the management of social media addiction in individuals which is decreasing the health of their lifestyle, attitude and family bonding.

To explain how abusive use of social media can increase the risk of psychological and behavioural problems.

DETAILED DESCRIPTION:
A sample of 150 individuals (male and female N=150) was recruited from different universities of Faisalabad for the purpose. A strategy of non-probability sampling of purposive technique was used for the recruitment of sample. The age range for the sample will be 18-22 as young adults and adults was targeted. Firstly individuals were screened out through social media addiction scale from which (n=60) participants were excluded because they did not meet the inclusion criteria of the study. Some participants left because lack of interest. After excluding (n=60) from the study rest of the participants (n=90) were randomized and allocated to experimental (n=45) and control group (n=45). After allocation of participants in the relevant group some participants were lost from the follow up from experimental (n=21) due to decline to participate and control group (n=20) due to lack of interest. Final analysis was conducted on experimental group and (n=24) control group (n=25) for the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals screened out through social media addiction scale will be used for the experimental study. Both male and female participants will be taken for the study. People with even mild score on social media addiction will be considered eligible for the study. Only people in the age range of 18-22 will be taken as participants in the study

Exclusion Criteria:

* Individuals not within the age range of 18-22 will not be taken as participants.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Social Media Addiction | 4 months
  Social media addiction scale was used to screen out the participants for eligibility assessment. Participants who will score high on the social media addiction scale will be enrolled
Insomnia severity index | 4
  This is 27 item scale which assess the quality of sleep.
Family relationship scale | 4
  Family relationship scale will be used to assess the person and family bonding and it will assess the impact of social media addiction

SECONDARY OUTCOMES:
Attitude and Belief Scale | 4
  This scale will assess the person general attitude and belief when he/she is using social media and being dependant

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas, PHD, Principal Investigator — Government College University Faisalabad
Locations (1):
- Qasir Abbas, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No